CLINICAL TRIAL: NCT06703606
Title: A PHASE 1B OPEN-LABEL NON-RANDOMIZED STUDY TO ASSESS THE SAFETY, PHARMACOKINETICS, AND PHARMACODYNAMICS OF MARSTACIMAB TREATMENT FOLLOWING THE DISCONTINUATION OF EMICIZUMAB THERAPY IN ADOLESCENT AND ADULT PARTICIPANTS WITH SEVERE HEMOPHILIA A WITHOUT INHIBITORS.
Brief Title: A Study to Learn About How Changing Therapy From Emicizumab to Marstacimab Affects People With the Severe Hemophilia A.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B7841014; NCT06703606 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2024-11-21; First posted 2024-11-25 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Severe Hemophilia A
Keywords: Hemophilia A; Severe Hemophilia A; Severe Hemophilia A Without Inhibitors
MeSH Terms: conditions — Hemophilia A | interventions — marstacimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MARSTACIMAB (Experimental): Marstacimab 150 mg subcutaneous (SC) once weekly (QW)
  Interventions: Drug: MARSTACIMAB

INTERVENTIONS:
Drug: MARSTACIMAB — Marstacimab 150 mg administered subcutaneous (SC) once weekly (QW)
  Other Names: PF-06741086

SUMMARY:
The purpose of the study is to learn about safety, how the body processes marstacimab and how it works in patients with severe hemophilia A without inhibitors. Hemophilia A is rare bleeding disorder where the blood doesn't clot normally. This causes a person to bleed a lot, even from a small cut.

These patients who are on emicizumab medicine for routine prophylaxis for at least 6 months, and desire to switch to marstacimab medicine. Inhibitors are antibodies that the immune system develops because it sees the infused clotting factor as a foreign substance that needs to be destroyed. Antibodies are proteins that eat up the activated factor before it has time to stop the bleeding. Prophylaxis are preventive medicines.

This study is seeking for participants:

* with severe Hemophilia A withouth inhibitors who are on emicizumab treatment for at least 6 months.
* must be 12 to less than 75 years old
* must have a body weight of at least 35 kilograms. The results from this study will serve as a guide to doctors and their hemophilia A patients who will change their medicines in the real-world clinical setting. Patients who can take part in the study will receive marstacimab medicine as weekly injections under the skin of 150 milligrams for 4 months. Study treatment with marstacimab will be initiated no earlier than 14 days after last dose of emicizumab. The study can last up to 6 months. The sponsor will provide marstacimab. Patients will continue their usual treatment with the infused clotting factor for their bleeds when taking part in the study. Roll-over into an optional study treatment extension period will be available to participants who wish to continue prophylaxis with marstacimab in countries where it is not commercially available.

DETAILED DESCRIPTION:
This is a non-randomized open-label study in approximately 10-15 adolescent and adult participants between ages 12 to <75 years with severe hemophilia A (defined as FVIII activity <1%) without inhibitors who are currently on treatment with emicizumab for ≥6 months. The study is designed to assess the safety and PK/PD during a 4-month treatment period with marstacimab 150 mg SC QW after a minimum 14-day wash-out period following discontinuation of emicizumab. Assessment of safety will be conducted by summarizing AEs and SAEs reported during the study, from the time each participant provides informed consent through and including a minimum of 28 calendar days after last dose of study intervention. Participants will continue to use their standard of care factor replacement for breakthrough bleeds during the course of the study. PK, PD, and ADA measurements will support the clinical safety data. The anticipated study duration for an individual participant is approximately 6 months. After completion of marstacimab treatment period participants will resume their standard of care prophylactic treatment after a 14-day wash-out period following the last dose of marstacimab. Roll-over into an optional study treatment extension period will be available to participants who wish to continue prophylaxis with marstacimab in countries where it is not commercially available.

ELIGIBILITY:
Inclusion Criteria:

1. Male and 12 to <75 years of age with a minimum body weight of 35 kg at the time of signing the informed consent.
2. Diagnosis of severe hemophilia A (FVIII activity <1%) without inhibitors.
3. On emicizumab therapy at a standard clinical dose for ≥6 months.

Exclusion Criteria:

1. Previous or current treatment for or history of coronary artery diseases, venous or arterial thrombosis, or ischemic disease.
2. Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
3. Known hemostatic defect other than hemophilia A.
4. Current use of any prohibited concomitant medication(s) or unwillingness or inability to use a required concomitant medication(s).
5. Previous administration of an investigational product (drug or vaccine) within 30 days or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer). Participation in studies of other investigational products (drug or vaccine) at any time during participation in this study.
6. Platelet count <100,000/μl or hemoglobin <10 g/dL.
7. Clinically significant renal or hepatic function abnormality based on laboratory results at screening, or known kidney or liver disease.
8. CD4 cell count ≤200/μl if HIV positive.
9. Screening 12-lead ECG that demonstrates clinically significant abnormalities that, in the opinion of the investigator, may affect participant safety or interpretation of study results.
10. Known planned surgical procedure.
11. Hypersensitivity or allergic reaction to hamster protein or other components of the study intervention.
12. Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor-delegate employees directly involved in the conduct of the study and their family members.

Ages: 12 Years to 74 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Adolescent and adult male patients
Enrollment: 15 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2027-05-05 (Estimated); Study Completion 2027-05-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of marstacimab-related adverse events (AEs) | Approximately 178 days: from the time the participant provides informed consent, through and including a minimum of 28 calendar days after last dose of study treatment
Incidence of marstacimab-related serious AEs (SAEs) | Approximately 178 days: from the time the participant provides informed consent, through and including a minimum of 28 calendar days after last dose of study treatment

SECONDARY OUTCOMES:
Plasma Concentration Versus Time of Marstacimab (Listings) | Day 1 up to day 135
Maximum Observed Plasma Concentration (Cmax) of Marstacimab | Day 1 up to day 135
Average Plasma Concentration (Cavg) of Marstacimab | Day 1 up to day 135
Minimum Observed Plasma Concentration (Cmin) | Day 1 up to day 135
Change from baseline in tissue factor pathway inhibitor (TFPI). | Baseline, Day 1 up to day 135
Change from baseline in prothrombin fragment 1+2 (PF 1+2) | Baseline, Day 1 up to day 135
Change from baseline in D-dimer | Baseline, Day 1 up to day 135
Change from baseline in TGA (thrombin generation assay). | Baseline, Day 1 up to day 135
Incidence of Anti-Drug Antibody (ADA) | Day 1 up to day 135
Incidence of clinically significant persistent neutralizing antibodies (NAb) | Day 1 up to day 135

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Orthopaedic Institute for Children, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7841014